CLINICAL TRIAL: NCT03000712
Title: Single-center, Randomized, Open Label, Negative-controlled Investigator Initiated Trial to Evaluate the Efficacy and Safety of Intra-articular Injection of ADMSC(Autologous Adipose Tissue Derived Mesenchymal Stem Cells) After High Tibial Osteotomy Compared to Negative Control in the Osteoarthritis Patients.
Brief Title: Investigator Initiated Trial to Evaluate the Efficacy and Safety of Intra-articular Injection of ADMSC Comared to Negative Control After High Tibial Osteotomy in the Osteoarthritis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R-Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTO-MSCs
Record Dates: First submitted 2016-12-18; First posted 2016-12-22 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2019-06

CONDITIONS: Degenerative Arthritis; Knee Osteoarthritis
Keywords: adipose tissue derived mesenchymal stem cell; osteoarthritis; degenerative arthritis; kyung hee university hospital; biostar; Rbio; Osteoarthritis, Knee; High tibial osteotomy; Joint Diseases
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous Adipose Tissue derived MSCs (Experimental): Biological: Autologous Adipose Tissue derived MSCs 1x10^8cells/3ml, 1 time injection(at 1week after high tibial osteotomy)
  Interventions: Biological: Autologous Adipose Tissue derived MSCs 1x10^8cells/3ml
- No treatment (No Intervention): No treatment (after high tibial osteotomy)

INTERVENTIONS:
Biological: Autologous Adipose Tissue derived MSCs 1x10^8cells/3ml — biological : Autologous Adipose Tissue derived MSCs 1x10^8cells/3ml drug: saline solution
  Other Names: JOINTSTEM
  Arms: Autologous Adipose Tissue derived MSCs

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intra-articular injection of autologous adipose tissue derived mesenchymal stem cells compared after high tibial osteotomy to negative control in the osteoarthritis patients

DETAILED DESCRIPTION:
In this clinical trial, the investigational product is administered intra-articularly at 1 week after high tibial osteotomy in a patient with degenerative arthritis of the medial side.

The investigational product is autologous adipose-derived mesenchymal stem cells. As it does not use allogenic tissue and is incubated without additional genetic modification or mechanical and chemical modification through differentiation, it is classified as 'autologous cell therapy' and is completely free of immunologic rejection.

It primarily aims to regenerate cartilage, to improve pain and joint function. The intra-articular injection of the investigational product is expected to stimulate the regeneration and growth of cartilage, and to innovatively improve pain and joint function with cartilage regeneration compared to high tibial osteotomy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must consent in writing to participate in the study by signing and dating an informed consent document
2. Patients who can communicate (exclusion of anyone who cannot understand the questionnaire)
3. between 20 years and 80 years of age
4. BMI≤30
5. Diagnosis of osteoarthritis by radiographic criteria of Kellgren and Lawrence grade 2-4
6. Diagnosis of osteoarthritis by ACR(American College of Rheumatology Criteria) Global functional criteria : There is the pain of the knee and radiographic osteophyte and at least one of the following (1) age >50 years (2) Less than 30 minutes of morning stiffness (3) The friction When moving weighted the knee
7. Patients who agree with contraception
8. Patients who agree to stop the existing osteoarthritis treatment and to get enough washout periods until medication time
9. Patients scheduled for High tibial osteotomy due to medial gonarthrosis

Exclusion Criteria:

1. patients with osteoporosis
2. Preparing for Pregnancy or Pregnant women or lactating mothers.
3. Patients with positive human immunodeficiency (HIV), hepatitis B (HBV), hepatitis C (HCV), venereal disease research laboratory(VDRL)
4. Patients with hypersensitivity to investigator product or investigational product component or those with a history
5. Patients who had participated in other clinical trials within 12 weeks prior to this study
6. Patients who received any drug by intra-articular injection for treatment within 2 months prior to this enrollment.
7. Patients who experienced as the knee joint cartilage and stem cell therapy or failure to treat
8. Patents who started or changed the physical therapy program established within 2 weeks before the start of the study or during the study(An established physical therapy program may continue for the duration of the trial, provided that it does not change in frequency and intensity)
9. Patents included in the following specific risk groups that may influence safety and efficacy assessments at the discretion of the investigator:: septic arthtritis, rheumatic disease, gout, recurrent pseudogout, paget disease, joint fracture, alcaptonuria, acromegaly, hemochromatosis, wilson's disease, primary osteochondrosis, hereditary disorder(ex: hyperkinesia), collagen gene abnormality ,etc
10. Patients who have clinically significant severe medical illnesses judged the principal investigator
11. Patients who have been diagnosed with malignancy within 5 years before screening (except for patients who were completely remissioned three years before screening criteria)
12. Patients who the principal investigator consider inappropriate for the clinical trial due to any other reasons
13. Patients who received concomitant contraindications and who have not passed the prescribed wash-out period before participating in the clinical trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
MRI scan | 24 months
  MRI perform to measure cartilage defect size change from baseline up to 27 weeks

SECONDARY OUTCOMES:
MRI scan | 15, 27 weeks, 18, 24 months
  MRI perform to measure cartilage defect size change from baseline up to 15 weeks
WOMAC score | 15, 27 weeks, 18, 24 months
  Change in WOMAC Total score from baseline up to 15, 27 weeks
WOMAC sub-scale | 15, 27 weeks, 18, 24 months
  Change in WOMAC sub-scale from baseline up to 15, 27 weeks
Kellgren & Lawrence grade | 15, 27 weeks, 18, 24 months
  Change in Kellgren & Lawrence grade from baseline up to 15, 27 weeks
EQ5D | 15, 27 weeks, 18, 24 months
  Change in the score of EQ-5D from baseline up to 15, 27 weeks
ROM | 15, 27 weeks, 18, 24 months
  change from baseline in knee flexion Range of Motion(ROM) at 15,27 weeks by physical examination
KOOS (Knee Injury & Osteoarthritis Outcome Score) | 15, 27 weeks, 18, 24 months
  Symptoms, pain and functionality of the knee joint will be evaluated via the Knee Injury and Osteoarthritis Outcome Score (KOOS)
PGIC(Patient Global Impression of Change) | 15, 27 weeks, 18, 24 months
  The percentage of subjects who were evaluated as improved at 15 weeks and 27 weeks in the patient global impression of change
PSQI(Pittsburgh Sleep Quality Index) | 15, 27 weeks, 18, 24 months
  Change in PSQI from baseline up to 15, 27 weeks
Biomarkers | 15, 27 weeks, 18, 24 months
  Change from baseline in Biomarkers up to 15, 27 weeks
Incidence of adverse reactions and characteristics associated with investigational product | 15, 27 weeks, 18, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: KANGIL KIM, M.D., Ph.D, Principal Investigator — KyungHee University Gangdong Hospital
Locations (1):
- KyungHee University Gangdong Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JH, Kim KI, Yoon WK, Song SJ, Jin W. Intra-articular Injection of Mesenchymal Stem Cells After High Tibial Osteotomy in Osteoarthritic Knee: Two-Year Follow-up of Randomized Control Trial. Stem Cells Transl Med. 2022 Jun 22;11(6):572-585. doi: 10.1093/stcltm/szac023. PMID 35674255